CLINICAL TRIAL: NCT07029126
Title: Improving the Perception of Stress and Mutuality in Caregivers (MI-DEAR Study) of Migraine Patients With Depressive Symptoms Treated With Fremanezumab: A Prospective Real-life Observational Study to Evaluate Whether Fremanezumab Reduces the Impact on Caregivers and Increases Couple Reciprocity
Brief Title: Improving the Perception of Stress and Mutuality in Caregivers (MI-DEAR Study) of Migraine Patients With Depressive Symptoms Treated With Fremanezumab: A Study to Evaluate Whether Fremanezumab Reduces the Impact on Caregivers and Increases Couple Reciprocity
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Other Study IDs: MI_DEAR
Record Dates: First submitted 2025-03-10; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2024-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PATIENTS: Adult male or female patients with diagnosis of migraine, with or without aura, or chronic migraine, according to the International Classification of Headaches (ICHD-3.)
  Interventions: Drug: Fremanezumab
- CAREGIVER: Adult subjects, male or female who are informal caregiver of enrolled migraine patients, defined as a person--spouse/partner, parent, child/child, sibling--who cares for the migraine patient, sharing the same household and performing various functions, from basic daily needs to socio-economic activities)

INTERVENTIONS:
Drug: Fremanezumab — subcutaneous injection 225 mg monthly or 675 mg quarterly
  Groups: PATIENTS

SUMMARY:
To evaluate the reduction of emotional burden (measured by Relative Stress Scale-RSS) of caregivers of migraine patients with Depressive Symptoms after 6 months after the first injection of fremanezumab.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS

* Adult patients, male or female
* Diagnosis of migraine, with or without aura, or chronic migraine, according to the International Classification of Headaches (ICHD-3.)
* Diagnosis of migraine with onset at an age of less than 50 years
* Depressive symptoms in patients defined as a Patient Health Questionnaire PHQ-9 scale score ≥5
* Complete details of migraine history and frequency of monthly migraine days in the past month
* clinical indication to start fremanezumab therapy to prevent migraine in patients naïve to monoclonal antibodies targeting the CGRP pathway
* In case of migraine preventive therapy and concomitant antidepressants, stability for at least 8 weeks prior to enrollment.
* Presence of a caregiver (see definition below) of the patient
* 80% compliance with diary and ability to complete the scale to provide written informed consent.

INFORMAL CAREGIVERS:

* Adult subjects, male or female.
* Informal caregiver is defined as a person--spouse/partner, parent, child/child, sibling--who cares for the migraine patient, sharing the same household and performing various functions, from basic daily needs to socio-economic activities)
* RSS score ≥ 1
* 80% compliance with completion scale ability to provide written informed consent

Exclusion Criteria:

Patients:

* Patients without a caregiver
* Contraindications or lack of indication to fremanezumab
* The patient has clinically significant hematological, cardiac, renal, endocrine, pulmonary, gastrointestinal, genitourinary, neurologic, hepatic, ocular disease, or complications of an infection, at the discretion of the investigator
* Patient with a clinical history of a severe or uncontrolled psychiatric disorder (bipolar disorders, schizophrenia, psychosis), at the discretion of the investigator, that would likely interfere with full participation in the study
* Patient participating in another study at the same time as enrollment in the current study

Informal Caregivers:

* History of migraine.
* History of major depressive disorder and severe or uncontrolled psychiatric disorder (bipolar disorders, schizophrenia, psychosis), at the discretion of the investigator, that would likely interfere with full participation in the study
* The caregiver has clinically significant hematological, cardiac, renal, endocrine, pulmonary, gastrointestinal, genitourinary, neurologic, hepatic, ocular disease, or complications of an infection at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of female and male patients aged >18 with a diagnosis of migraine with and without aura (as defined by the International Classification of Headache Disorders, ICHD-3)15. Patients must have been diagnosed with migraine at least 12 months before the baseline visit, and the diagnosis of migraine will be confirmed via a review of the medical chart and of a 4-week headache diary before the baseline visit.
  Only patients with an indication to start a new preventive medication with fremanezumab and their caregivers will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
CHANGE in caregiver stress | from baseline to evaluation at 6 months after fremanezumab therapy
  Change in Relative Stress Scale (RSS) scores in caregivers (range 15-60, where 15 is no stress and 60 maximum stress)

SECONDARY OUTCOMES:
CHANGE IN RECIPROCITY | from baseline to the evaluation after 6 months of therapy with fremanezumab
  To evaluate an increase in reciprocity within the mutuality scale in the caregiver/ migraine patient dyad after 6 months from the first injection of fremanezumab.
  Reciprocity represents the mean value of the response to questions 5, 6, 10, 13, and 15 of the mutuality scale (raging from 0, lower reciprocity, to 4 higher reciprocity)
CORRELATION BETWEEN CHANGE IN patient depression and caregiver stress | from baseline to 6 months after fremanezumab therapy
  to evaluate whether the change in depression (Patient Health Questionnaire. PHQ-9 scores, range 0-27; higher scores indicate more severe depression) in migraine patients 6 months after starting fremanezumab is associated with the change of stress (Relative Stress Scale) in caregivers.
CORRELATION BETWEEN THE CHANGES IN DEPRESSION AND RECIPROCITY SCALE SCORES | from baseline to 6 months after therapy with fremanezumab
  To evaluate whether the CHANGE in depressive (PHQ-9 SCALE) and anxiety (STAY SCALE) symptoms in migraine patients 6 months after starting fremanezumab is associated with the change in reciprocity (MUTUALITY SCALE) between patient and caregiver
PATIENT ANXIETY AND CAREGIVER STRESS | from baseline to 6 months after fremanezumab therapy
  to evaluate whether the change in anxiety (STATE-TRAIT ANXIETY INVENTORY STAY, range 20-80, from 40 points to higher scores indicate anxiety) symptoms in migraine patients 6 months after starting fremanezumab is associated with the change of stress (Relative Stress Scale) in caregivers
PATIENT DISABILTY AMD CAREGIVER STRESS | from baseline to 6 months after fremanezumab therapy
  to evaluate whether the change in anxiety disability (MiGRAINE DISABILITY ASSESSMENT MIDAS raging from 0 to 270, higher scores indicate greater disability) in migraine patients 6 months after starting fremanezumab is associated with the change of stress (Relative Stress Scale) in caregivers

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Italy
  - Ospedali Riuniti "Umberto I"- GM LANCISI G.SALESI, Ancona
  - PO Avezzano "S.Filippo e Nicola", Avezzano
  - Clinica Neurologica "L. Amaducci" Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, Bari
  - IRCCS Istituto Scienze Neurologiche, Bologna
  - ASST Spedali Civili Brescia, Brescia
  - Fondazione IRCCS Istituto Neurologico "Carlo Besta, Milan
  - Dipartimento delle scienze avanzate mediche e chirurgiche, Università della Campania "Luigi Vanvitelli, Naples
  - IRCCS San Raffaele Pisana, Rome
  - Ospedale Fabenefratelli- San Pietro, Rome

IPD SHARING:
Plan to Share IPD: No